CLINICAL TRIAL: NCT05772455
Title: A Phase I, Open-label, Dose-escalation Study of the Safety, Pharmacokinetics and Efficacy of the XZB-0004 in Patients With Solid Tumours
Brief Title: A Study of XZB-0004 in Patients With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZB-0004-1001
Record Dates: First submitted 2023-02-20; First posted 2023-03-16 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor; NSCLC
Keywords: XZB-0004; AXL inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XZB-0004 (Experimental)
  Interventions: Drug: XZB-0004

INTERVENTIONS:
Drug: XZB-0004 — Part 1a: 100mg BID, 150mg BID, and 200mg BID of XZB-0004 are planned to be evaluated, and the possibility of exploring higher or lower doses is not ruled out. Continuous administration of XZB-0004 for 21 days is a treatment cycle. Part 1b: XZB-0004 in combination with Penpulimab in subjects with advanced NSCLC or solid tumors, starting at a dose level down from the RP2D of XZB-0004 monotherapy- cohort 1: Advanced or metastatic NSCLC with advanced disease progression after treatment with PD-1 or PD-L1 inhibitors; cohort 2: Advanced or metastatic NSCLC with advanced disease progression after platinum-containing chemotherapy without prior use of any immunocheckpoint inhibitors; cohort3: Advanced or metastatic solid tumors that cannot be radically cured by surgery or local therapy, including but not limited to urothelial carcinoma, melanoma, etc. Subjects had disease progression since last antitumor therapy, no availability or intolerance or refusal of standard therapy.

SUMMARY:
XZB-0004 is a novel and potent small molecule inhibitor of receptor tyrosine kinase AXL.

This is an open-label, multicentre phase I study of XZB-0004 in patients with solid tumors. Part 1 is a dose-escalation study to evaluate the safety, pharmacokinetic (PK), and pharmacodynamic profile of XZB-0004, and then to identify a safe and pharmacologically active dose for evaluation in subsequent cohorts or clinical studies. Part 2 is a study to evaluate the efficacy and safety of XZB-0004 combined with Penpulimab in patients with NSCLC or advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed informed consent before any trial related activities.
2. Be 18 years of age or older and less than 75 years at the time of signing the informed consent.
3. Part 1: Have a histologically or cytologically confirmed diagnosis of a solid tumour malignancy; Part 2：Have a histologically or cytologically confirmed diagnosis of a NSCLC or solid tumour malignancy.
4. Have evaluable (for Part 1) or measurable (for Part 2) disease as the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
5. Have a performance status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
6. Have adequate organ function.
7. Have recovered to ≤ grade 1 or Meet the requirements of the study from the effects of any prior cancer therapy, except for alopecia; irreversible neuropathy should have recovered to ≤ grade 2.
8. Have a life expectancy greater than 3 months.
9. Eligible patients (male and female) who are fertile must agree to at least use a reliable contraceptive method with partner.
10. Willingness to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Previous use of AXL inhibitors and immunotherapy was consistent with protocol requirements.
2. Received anti-tumor therapy such as chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy or other therapy within 4 weeks prior to the first dose of the investigational drug.
3. Received other unmarketed investigational drugs or treatments within 4 weeks or 5 times the elimination half-life prior to the first dose of the investigational drug.
4. Treatment with systemic glucocorticoids (prednisone > 10mg per day or equivalent) or other immunosuppressive agents within 14 days before the first dose of a trial drug.
5. Inability to swallow, intestinal obstruction or other factors that affect the taking and absorption of the drug.
6. Patient with heart function impaired or clinically significant heart disease.
7. Any condition or illness that, in the opinion of the Investigator, would interfere with the evaluation of the safety of the study drug.
8. History of immune deficiencies, including positive HIV antibody tests.
9. Patient is in the active stage of HBV or HCV.
10. History of solid organ transplant or bone marrow transplant.
11. Any other malignant tumor has been diagnosed within 5 years.
12. Has known Primary tumor of the central nervous system or central nervous system metastase.
13. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage were present within 4 weeks before the first dose of the trial drug.
14. Subjects with psychiatric disorders that may affect trial compliance.
15. history of Alcoholism or drug abuse.
16. Pregnant or breastfeeding.
17. The researchers considered that there were some cases that were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (for Part 1a) | Up to 3 weeks
  Determine MTD of XZB-0004
Recommended phase 2 dose (RP2D）(for Part 1a) | Up to 3 weeks
  Determine RP2D of XZB-0004
Overall Response Rate (ORR) (for Part 1b) | Up to 2-3 years
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Pharmakinetic parameter - AUC0-t (for Part 1a and Part 1b) | Up to 63 days
  To determine AUC0-t of XZB-0004
Pharmakinetic parameter - AUC0-∞ (for Part 1a and Part 1b) | Up to 63 days
  To determine AUC0-∞ of XZB-0004
Pharmakinetic parameter - Cmax (for Part 1a and Part 1b) | Up to 63 days
  To determine Cmax of XZB-0004
Pharmakinetic parameter - Tmax (for Part 1a and Part 1b) | Up to 63 days
  To determine Tmax of XZB-0004
Pharmakinetic parameter - t½ (for Part 1a and Part 1b) | Up to 63 days
  To determine t½ of XZB-0004
Pharmakinetic parameter - CL/F (for Part 1a and Part 1b) | Up to 63 days
  To determine CL/F of XZB-0004
Pharmakinetic parameter - Vz/F (for Part 1a and Part 1b) | Up to 63 days
  To determine Vz/F of XZB-0004
Overall Response Rate (ORR) (for Part 1a) | Up to 2-3 years
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression free survival (PFS) (for Part 1a and Part 1b) | Up to 2-3 years
  PFS is defined as the time from the date of first dose of XZB-0004 till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Duration of response (DOR) (for Part 1a and Part 1b) | Up to 2-3 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) (for Part 1a and Part 1b) | Up to 2-3 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1.
Overall survival (OS) (for Part 1a and Part 1b) | Up to 2-3 years
  OS is the time from the date of first dose of XZB-0004 to death due to any cause.
Incidence and severity of adverse events (AEs)(for Part 1b) | Up to 2-3 years
  An adverse event (AE) is any untoward medical occurrence or the deterioration of existing medical event in a clinical study subject administered an investigational drug, which does not necessarily have an unequivocal causal relationship with the investigational product.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China